CLINICAL TRIAL: NCT04288089
Title: An Open-Label Multicenter Phase 1b Study of H3B-6545 in Combination With Palbociclib in Women With Advanced or Metastatic Estrogen Receptor-Positive HER2-Negative Breast Cancer
Brief Title: A Study of H3B-6545 in Combination With Palbociclib in Women With Advanced or Metastatic Estrogen Receptor-Positive Human Epidermal Growth Factor Receptor-2 (HER2)-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H3B-6545-G000-102; 2019-004622-17 (EudraCT Number)
Record Dates: First submitted 2020-02-26; First posted 2020-02-27 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Receptors, Estrogen; Genes, Erbb-2; Breast Neoplasms
Keywords: H3B-6545; Palbociclib; Metastatic Estrogen Receptor-Positive; HER2-Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; H3B-6545

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Palbociclib + H3B-6545 (Dose Escalation and Dose Expansion) (Experimental): Participants will receive Palbociclib 75, 100, 125 milligram (mg) capsules or tablets, orally, once daily from Days 1 to 21 followed by 7 days off treatment in 28-day cycles along with H3B-6545 150, 300, 450 mg capsules or tablets, orally, once daily from Days 1 to 28 in 28-day cycles in dose escalation part. Based on MTD or RP2D determined for H3B-6545 in combination with palbociclib in dose escalation part, participants will continue to receive study treatment in dose expansion part until PD, development of unacceptable toxicity, or withdrawal of consent (up to 24 months).
  Interventions: Drug: Palbociclib (75, 100, 125 milligram [mg]); Drug: H3B-6545 (150, 300, 450 mg)

INTERVENTIONS:
Drug: Palbociclib (75, 100, 125 milligram [mg]) — Palbociclib orally, once daily (QD).
Drug: H3B-6545 (150, 300, 450 mg) — H3B-6545 orally, QD.

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of H3B-6545 and palbociclib when administered in combination in order to determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of this combination in women with advanced or metastatic estrogen receptor-positive (ER+) HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. ER+ HER2- locally advanced, recurrent, or metastatic breast cancer, as per local laboratory
2. Prior therapy in the advanced/metastatic setting
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Has adequate bone marrow and organ function

Exclusion Criteria:

1. Uncontrolled significant active infections
2. Major surgery or other locoregional treatment within 4 weeks before the 1st dose of study drug
3. Inability to take oral medication or presence of malabsorption
4. Active cardiac disease or a history of cardiac dysfunction
5. Evidence of ongoing Alcohol or Drug Abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Florida Cancer Specialists South - SCRI - PPDS, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Tennessee Oncology, PLLC - SCRI - PPDS, Nashville, Tennessee
- United Kingdom (3):
  - Royal Marsden NHS Foundation Trust, London
  - Sarah Cannon Research Institute UK - SCRI, London
  - Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Furman C, Puyang X, Zhang Z, Wu ZJ, Banka D, Aithal KB, Albacker LA, Hao MH, Irwin S, Kim A, Montesion M, Moriarty AD, Murugesan K, Nguyen TV, Rimkunas V, Sahmoud T, Wick MJ, Yao S, Zhang X, Zeng H, Vaillancourt FH, Bolduc DM, Larsen N, Zheng GZ, Prajapati S, Zhu P, Korpal M. Covalent ERalpha Antagonist H3B-6545 Demonstrates Encouraging Preclinical Activity in Therapy-Resistant Breast Cancer. Mol Cancer Ther. 2022 Jun 1;21(6):890-902. doi: 10.1158/1535-7163.MCT-21-0378. PMID 35642432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in the United States and the United Kingdom from 1 April 2020 to 16 September 2022.
Pre-assignment Details: This study was planned to be conducted in two parts: Dose Escalation and Dose Expansion. In the Dose Escalation part, a total of 31 participants were enrolled and received the study treatment. However, no participants were enrolled in the Dose Expansion part. In this result summary, data has been reported for dose escalation part only and up to primary completion date (16 September 2022). This study is ongoing and will be updated with final results after study completion.
Groups:
- H3B-6545 300 mg + Palbociclib 100 mg: Participants received palbociclib 100 milligram (mg) capsule, orally, once daily (QD) from Days 1 to 21 followed by H3B-6545 300 mg capsule, orally, QD from Days 9 to 28 in Cycle1. In all 28 days subsequent cycles, palbociclib was administered on Days 1 to 21, and H3B-6545 was administered on Days 1 to 28 until disease progression, development of unacceptable toxicity, or withdrawal of consent.
- H3B-6545 300 mg + Palbociclib 125 mg: Participants received palbociclib 125 mg capsule, orally, QD from Days 1 to 21 followed by H3B-6545 300 mg capsule, orally, QD from Days 9 to 28 in Cycle1. In all 28 days subsequent cycles, palbociclib was administered on Days 1 to 21, and H3B-6545 was administered on Days 1 to 28 until disease progression, development of unacceptable toxicity, or withdrawal of consent.
- H3B-6545 450 mg + Palbociclib 125 mg: Participants received palbociclib 125 mg capsule, orally, QD from Days 1 to 21 followed by H3B-6545 450 mg capsule, orally, QD from Days 9 to 28 in Cycle1. In all 28 days subsequent cycles, palbociclib was administered on Days 1 to 21, and H3B-6545 was administered on Days 1 to 28 until disease progression, development of unacceptable toxicity, or withdrawal of consent.
- H3B-6545 450 mg + Palbociclib 100: Participants received palbociclib 100 mg capsule, orally, QD from Days 1 to 21 followed by H3B-6545 450 mg capsule, orally, QD from Days 9 to 28 in Cycle1. In all 28 days subsequent cycles, palbociclib was administered on Days 1 to 21, and H3B-6545 was administered on Days 1 to 28 until disease progression, development of unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | H3B-6545 300 mg + Palbociclib 100 mg | H3B-6545 300 mg + Palbociclib 125 mg | H3B-6545 450 mg + Palbociclib 125 mg | H3B-6545 450 mg + Palbociclib 100
Started | 7 | 8 | 8 | 8
Completed | 5 | 7 | 7 | 4
Not Completed | 2 | 1 | 1 | 4
Not completed — Ongoing Treatment | 2 | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | H3B-6545 300 mg + Palbociclib 100 mg | H3B-6545 300 mg + Palbociclib 125 mg | H3B-6545 450 mg + Palbociclib 125 mg | H3B-6545 450 mg + Palbociclib 100 | Total
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (7.76) | 51.9 (15.61) | 56.0 (4.96) | 59.1 (14.53) | 57.2 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 8 | 8 | 31
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 8 | 8 | 6 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 6 | 8 | 8 | 5 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of H3B-6545 and Palbociclib
Description: The MTD was defined as the highest dose at which no more than 1 of 6 participants experienced a Dose-Limiting Toxicity (DLT) in the dose cohort. DLT was graded as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. DLTs were defined as the following events that occurred in Cycle 1, for which a causal relationship with the study drug could not be ruled out: febrile neutropenia; Grade 4 neutropenia that was not resolved within 7 days; Grade 4 thrombocytopenia; Grade 3 thrombocytopenia lasting greater than (>) 7 days or associated with clinically significant bleeding; Grade 4 vomiting and diarrhea; Grade 3 vomiting and diarrhea lasting > 72 hours despite treatment; Grade 4 electrolyte abnormality or Grade 3 abnormality lasting > 24 hours; Grade 3 or 4 serum creatinine or bilirubin increase; Grade 4 biochemistry or Grade 3 lasting > 7 days; Grade 4 or Grade 3 or intolerable grade 2 toxicities of any non-hematologic adverse event.
Time Frame: Cycle 1 (Cycle length = 28 Days)
Population: The Dose Evaluable Set (DES) included all participants who were evaluated for DLTs in dose escalation part.
Measure: Number; unit: milligram
Groups:
- All Participants: Participants received palbociclib (100 mg, 125 mg) from Days 1 to 21 followed by H3B-6545 (300 mg, 450 mg), from Days 9 to 28 in Cycle1. In all 28 days subsequent cycles, palbociclib was administered on Days 1 to 21, and H3B-6545 on Days 1 to 28 until disease progression, development of unacceptable toxicity, or withdrawal of consent.
Arm/Group | All Participants
Number analyzed (Participants) | 28
milligram
  Palbociclib | 125
  H3B-6545 | 300

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAE was defined as an adverse event (AE) with an onset that had occurred after receiving study drug. An AE was defined as any untoward medical occurrence in a participants or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. A serious adverse event (SAE) was defined as any AE if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect. Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: From first dose up to 28 days after the last dose of study drug (up to Month 48)
Reporting Status: Not Posted, anticipated posting 2026-03

3. Secondary Outcome: AUC(0-t): Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Point for Palbociclib and H3B-6545
Description: Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: Dose Escalation Part: Cycle 1 Days 8, 21 and 28: 0-24 hours postdose; Dose Expansion Part: Cycle 1 Day 21: 0-24 hours postdose (Each Cycle length=28 days)
Reporting Status: Not Posted, anticipated posting 2026-03

4. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Palbociclib and H3B-6545
Description: Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2026-03

5. Secondary Outcome: Tmax: Time to Reach the Cmax for Palbociclib and H3B-6545
Description: Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: C24: Plasma Concentration at 24 Hour Post-dose for Palbociclib and H3B-6545
Description: Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2026-03

7. Secondary Outcome: Ratio of Pharmacokinetic (PK) Cmax Parameter Estimates Between Day 21 (Palbociclib) and Day 8 (Palbociclib)
Description: Ratio of palbociclib Cmax Day 21/Day 8, is the ratio of palbociclib exposure on Day 21 and palbociclib exposure on Day 8. Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: Dose Escalation Part: Cycle 1 Days 8 and 21: 0-24 hours postdose
Reporting Status: Not Posted, anticipated posting 2026-03

8. Secondary Outcome: Ratio of PK AUC24 Parameter Estimates Between Day 21 (Palbociclib) and Day 8 (Palbociclib)
Description: Ratio of palbociclib AUC24 Day 21/Day 8, is the ratio of palbociclib exposure on Day 21 and palbociclib exposure on Day 8. Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: Dose Escalation Part: Cycle 1 Days 8 and 21: 0-24 hours postdose; Dose Expansion Part: Cycle 1 Day 21: 0-24 hours postdose (Each Cycle length=28 days)
Reporting Status: Not Posted, anticipated posting 2026-03

9. Secondary Outcome: Ratio of PK C24 Parameter Estimates Between Day 21 (Palbociclib) and Day 8 (Palbociclib)
Description: Ratio of palbociclib C24 Day 21/Day 8, is the ratio of palbociclib exposure on Day 21 and palbociclib exposure on Day 8. Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: as for outcome 8
Reporting Status: Not Posted, anticipated posting 2026-03

10. Secondary Outcome: Ratio of PK Cmax Parameter Estimates Between Day 21 (H3B-6545) and Day 28 (H3B-6545)
Description: Ratio of palbociclib Cmax Day 21/Day 28, is the ratio of H3B-6545 exposure on Day 21 and H3B-6545 exposure on Day 28. Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: Dose Escalation Part: Cycle 1 Days 21 and 28: 0-24 hours postdose; Dose Expansion Part: Cycle 1 Day 21: 0-24 hours postdose (Each Cycle length=28 days)
Reporting Status: Not Posted, anticipated posting 2026-03

11. Secondary Outcome: Ratio of PK AUC24 Parameter Estimates Between Day 21 (H3B-6545) and Day 28 (H3B-6545)
Description: Ratio of H3B-6545 AUC24 Day 21/Day 28, is the ratio of H3B-6545 exposure on Day 21 and H3B-6545 exposure on Day 28. Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: as for outcome 10
Reporting Status: Not Posted, anticipated posting 2026-03

12. Secondary Outcome: Ratio of PK C24 Parameter Estimates Between Day 21 (H3B-6545) and Day 28 (H3B-6545)
Description: Ratio of H3B-6545 C24 Day 21/Day 28, is the ratio of H3B-6545 exposure on Day 21 and H3B-6545 exposure on Day 28. Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: as for outcome 10
Reporting Status: Not Posted, anticipated posting 2026-03

13. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants achieving a best overall response (BOR) of confirmed partial response (PR) or complete response (CR). The ORR will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: From first dose of study drug up to Month 48
Reporting Status: Not Posted, anticipated posting 2026-03

14. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the date of the first documented CR/PR until the first documentation of disease progression (PD) or death, whichever comes first. The DoR will be assessed according to RECIST version 1.1. Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: From the date of first documented CR/PR until the PD or death, whichever occurs first (up to Month 48)
Reporting Status: Not Posted, anticipated posting 2026-03

15. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants with BOR of PR, CR, or durable stable disease (SD) (duration of SD greater than or equal to 23 weeks). Duration of SD is defined as the time from the date of first dose to the date of the first documentation of disease progression or death, whichever occurs first. It will be calculated for participants whose BOR is SD. The CBR will be assessed according to RECIST version 1.1. Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: From the first dose of study drug until disease progression or death, whichever occurs first (up to Month 48)
Reporting Status: Not Posted, anticipated posting 2026-03

16. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from the first dose date to the date of the first documentation of PD or death (whichever occurs first). Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: From first dose of study drug until first documentation of PD or death, whichever occurs first (up to Month 48)
Reporting Status: Not Posted, anticipated posting 2026-03

17. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first dose date to the date of death from any cause. Analysis is not final for this outcome measure, and complete data will be posted at study completion date.
Time Frame: From the date of first dose to the date of death from any cause (up to Month 48)
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: First dose of study drug to approximately up to 29 months
Arm/Group | H3B-6545 300 mg + Palbociclib 100 mg | H3B-6545 300 mg + Palbociclib 125 mg | H3B-6545 450 mg + Palbociclib 125 mg | H3B-6545 450 mg + Palbociclib 100
All-Cause Mortality (participants affected / at risk) | 3/7 | 3/8 | 4/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/7 | 2/8 | 3/8 | 3/8
Other Adverse Events (participants affected / at risk) | 7/7 | 7/8 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | H3B-6545 300 mg + Palbociclib 100 mg (N=7) | H3B-6545 300 mg + Palbociclib 125 mg (N=8) | H3B-6545 450 mg + Palbociclib 125 mg (N=8) | H3B-6545 450 mg + Palbociclib 100 (N=8)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | H3B-6545 300 mg + Palbociclib 100 mg (N=7) | H3B-6545 300 mg + Palbociclib 125 mg (N=8) | H3B-6545 450 mg + Palbociclib 125 mg (N=8) | H3B-6545 450 mg + Palbociclib 100 (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 4 | 7
Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 2 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 5 | 5 | 4 | 7
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 4 | 4
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4 | 2
Chest discomfort (General disorders) | 0 | 0 | 1 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 6 | 2
Malaise (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 3 | 1 | 2
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 3 | 2
Amylase increased (Investigations) | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1 | 3
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 0
Lipase increased (Investigations) | 1 | 0 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 4 | 5
Oxygen saturation decreased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 2 | 2 | 3
Serum ferritin increased (Investigations) | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 2 | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Allodynia (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT04288089/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT04288089/SAP_001.pdf